CLINICAL TRIAL: NCT02744703
Title: Professor, Ege University Faculty of Dentistry
Brief Title: Effect of Caffeic Acid Phenethyl Ester as a Matrix Metalloproteinase Inhibitor: Randomized Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Mine Dundar Comlekoglu, Professor, Ege University Faculty of Dentistry, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 04.10.2012; no:12-8/6
Record Dates: First submitted 2016-04-03; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Matrix Metalloproteinase Inhibitors; Composite Resins
MeSH Terms: interventions — Adhesives

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- self-etch adhesive (Active Comparator): application of self-etch adhesive on cavities.
  Interventions: Drug: self-etch adhesive
- CAPE-S (Experimental): CAPE before self-etch adhesive
  Interventions: Drug: CAPE-S
- total-etch adhesive (Active Comparator): total-etch adhesive on cavities.
  Interventions: Drug: total-etch adhesive
- CAPE-T (Experimental): CAPE before total-etch adhesive application
  Interventions: Drug: CAPE-T

INTERVENTIONS:
Drug: total-etch adhesive — comparator use of total-etch adhesive
  Other Names: adhesive
  Arms: total-etch adhesive
Drug: CAPE-T — experimental group
  Other Names: CAPE solution
  Arms: CAPE-T
Drug: self-etch adhesive — comparator use of total-etch adhesive
  Other Names: adhesive
  Arms: self-etch adhesive
Drug: CAPE-S — experimental group
  Other Names: CAPE solution
  Arms: CAPE-S

SUMMARY:
Matrix metalloproteinases (MMPs); activated by the application of adhesive systems on dentin cause degradation of the collagen proteins and loss of bond strength in adhesive restorations. Caffeic acid phenethyl ester (CAPE) showed inhibitory activities on dentinal MMPs. It is hypothesised that dentin pretreatment with CAPE, as an MMP inhibitor, would be beneficial for the bonding of resin material and tooth substrate over the course of time. This study evaluated the effect of 5 % CAPE pretreatment on the microtensile bond strength of a nanohybrid resin restoration applied with total-etch or self-etch adhesive systems on 10 patients (12-18 yrs). Two standard cavities (3 x 3 x 4 mm) prepared on the occlusal surfaces of one of the two premolar teeth in each patient were randomly assigned into four treatment groups (n=10); 5% CAPE pretreatment and total-etch adhesive (TC), Total-etch adhesive (control) (T), 5% CAPE pretreatment and self-etch adhesive (SC), Self-etch adhesive (control) (S) followed by restoration and 3 months of intra-oral functioning. After teeth extraction, the specimens were stored in distilled water+thymol solution at 4°C to inhibit microbial growth and used in one week period. Dentin-composite sticks were obtained from each restoration for µTBS tests and scanning electron microscopy (SEM) evaluation. Failure mode analysis was performed microscopically. Data were analysed statistically using Repeated Measure ANOVA (p < 0.05). Dentin pretreatment with CAPE solution (5%) for 60 seconds significantly increased the composite resin restorations' bond strengths to dentin applied with either total-etch or self-etch adhesive system. Thus it can be used as an MMP inhibitor prior to the the resin restorations. However further long term clinical studies are needed to support the use of CAPE pretreatment along with self-etch and total-etch adhesive systems.

DETAILED DESCRIPTION:
The aim of the present study was to evaluate the effect of caffeic acid phenethyl ester (CAPE) pretreatment used as matrix metalloproteinase (MMP) inhibitor on microtensile bond strength (µTBS) of nanohybrid resin restorations applied with total-etch or self-etch adhesive systems. A total of 10 patients aged between 12 and 18 years old (4 males, 6 females, mean age:15) received 40 composite restorations. The patients who had contralateral pairs of caries-free premolars which were planned to be extracted for orthodontic treatment were enrolled in the study. This study was performed with a protocol approved by the Ethical Committee for Clinical Studies, Faculty of Medicine, University of Ege, Izmir, Turkey (04.10.2012; no:12-8/6). The treatments were performed after the informed consents were received both from the parents and the patients. Included teeth were in function and no anomalies were found neither in teeth nor in occlusion. Two standard cavities (3 x 3 x 4 mm) with continuous enamel cavosurface margins were prepared on the occlusal surfaces of each premolar tooth.Totally four cavities in each patient were randomly assigned into four treatment groups (n=10); Group TC: CAPE and total-etch adhesive (Syntac; Ivoclar Vivadent AG), Group T: Total-etch adhesive (control), Group SC: CAPE and self-etch adhesive (AdheSE; Ivoclar Vivadent AG), Group S: Self-etch adhesive (control). All cavities were restored incrementally with a nano-filled hybrid composite resin (Tetric-N-Ceram, Ivoclar Vivadent AG) in which polymerization in each layer was performed for 40 seconds with a light-curing unit (BluePhase Ivoclar Vivadent AG) exceeding an energy output of 500mw/sec.

ELIGIBILITY:
Inclusion Criteria:I

* Occlusally functioning teeth without any anomalies
* Good oral hygiene
* No systemical disorders
* No periodontal diseases
* No allergic reactions to the dental materials

Exclusion Criteria:

* Patients not eligible for premolar teeth extraction for orthodontic treatment
* Poor oral hygiene
* Non-functioning premolar teeth to be included
* Patients having systemical disorders, periodontal diseases or allergic reactions to dental materials

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Determination of structural integrity of hybrid layer in forty restorations on 10 patients using scanning electron microscopy after application of different adhesive strategies and a matrix metalloproteinase inhibitor. | 2 years

IPD SHARING:
Plan to Share IPD: Undecided